CLINICAL TRIAL: NCT04992026
Title: A Randomized, Controlled, Multi-Center Clinical Trial to Evaluate the Efficacy and Safety of Prostatectomy for Castration-Naive Oligometastatic Prostate Cancer
Brief Title: The Efficacy and Safety of Prostatectomy for Castration-Naive Oligometastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other); The First People's Hospital of Changzhou (Other); The First Affiliated Hospital of Soochow University (Other); Wuxi People's Hospital (Other); The Affiliated Hospital of Nantong University (Unknown); The Affiliated Hospital of Yangzhou University (Unknown)
Responsible Party: Principal Investigator, Hongqian Guo, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-108
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Prostatectomy; Oligometastatic Prostate Cancer; Abiraterone
MeSH Terms: interventions — Prednisone; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADT plus abiraterone + surgery (Experimental): After 6 cycles of first-line treatment (Androgen deprivation therapy + abiraterone acetate along with prednisone) , patients will receive robot assisted laparoscopic prostatectomy + enlarged pelvic lymph node dissection (ePLND) within 9 months of being diagnosed. The ADT+abiraterone treatment will be maintained after surgery.
  Interventions: Procedure: robot assisted laparoscopic prostatectomy + enlarged pelvic lymph node dissection; Drug: 1.Abiraterone Acetate Tablets; Drug: Prednisone Acetate Tablets; Drug: Luteinizing Hormone-Releasing Hormone Analog
- ADT plus abiraterone (Active Comparator): Patients will be only treated with Androgen deprivation therapy + abiraterone acetate along with prednisone. Prostatectomy won't be performed.
  Interventions: Drug: 1.Abiraterone Acetate Tablets; Drug: Prednisone Acetate Tablets; Drug: Luteinizing Hormone-Releasing Hormone Analog

INTERVENTIONS:
Procedure: robot assisted laparoscopic prostatectomy + enlarged pelvic lymph node dissection — Robot assisted laparoscopic prostatectomy + enlarged pelvic lymph node dissection will be performed.
  Arms: ADT plus abiraterone + surgery
Drug: 1.Abiraterone Acetate Tablets — 1000mg(4 tablets, 250mg per tablet) daily for 6 cycles
Drug: Prednisone Acetate Tablets — 5 mg oral low dose prednisone taken along with Abiraterone Acetate Tablets
Drug: Luteinizing Hormone-Releasing Hormone Analog — Hypodermic injection of Luteinizing Hormone-Releasing Hormone Analog every 4 weeks including goserelin, leuprolide, triptorelin ect.

SUMMARY:
This randomized, controlled, multi-center clinical trial aims to evaluate the efficacy and safety of prostatectomy for castration-Naive oligometastatic prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 40 and ≤75 years of age.
* All patients must have a histologically or cytologically diagnosis of prostate cancer.
* All patients must have been diagnosed oligometastatic prostate cancer which meet the following criteria. (1) ≤5 metastatic lesions are found by imaging examination (2)No visceral metastasis was found (3) The diameter of a single lesion ≤5cm or the surface area ≤250cm2.
* Patients previously treated with surgical castration or androgen deprivation therapy must maintain a testosterone level of <50ng/dl or <1.7nmol/L during treatment. Also the treatment duration should be less than 9 months. Patients were previously treated with at least 6 cycles of abiraterone.
* PSA<2ng/ml before enrollment.
* There was no PSA progression or radiographic progression during previous treatment.
* Primary lesion must be eligible for radical prostatectomy based on random radiographic assessment. ( Preoperative clinical staging <T4 or achievable complete resection agreed by experienced surgeons is deemed as eligible for radical prostatectomy)
* Eastern Cooperative Oncology Group (ECOG) physical condition score ≤ 1.
* Patients must have adequate hematologic function, within 28 days prior to registration as evidenced by: white blood cell (WBC) ≥ 4.0 × 109 /L, platelets≥ 100 × 109 / L, hemoglobin ≥ 9g / dL, and international normalized ratio (INR) < 1.5.
* Patients must have adequate hepatic function, within 28 days prior to registration, as evidenced by: total bilirubin (TBIL)≤1.5 x upper limit of normal (ULN),and SGOT (AST) and SGPT (ALT) ≤ 2.5 x ULN.
* Patients must have adequate renal function, within 28 days prior toregistration, as evidenced by serum creatinine ≤2×ULN
* Patients must participate voluntarily and sign an informed consent form(ICF), indicating that they understand the purpose and required procedures of the study, and are willing to participate in. Patients must be willing to obey the prohibitions and restrictions specified in the research protocol.

Exclusion Criteria:

* Patients with neuroendocrine, small cell, or signet ring cell histological features are not eligible.
* Patients with visceral metastasis or more than 5 metastatic lesions are excluded.
* Patients were diagnosed metastatic castration-naive prostate cancer for more than 9 months or showed biochemical or radiographic progression before enrollment.
* Patients with unresectable primary lesion before enrollment based on CT/MRI.
* Patients received local treatments such as pre-focal treatment, radiotherapy and palliative endoscopic resection.
* Patients with severe or uncontrolled concurrent infections are not eligible.
* Patients must not have New York Heart Association Class III or IV congestive heart failure at the time of screening. Patients must not have any thromboembolic event, unstable angina pectoris, myocardial infarction within 6 months prior to registration.
* Patients must not have uncontrolled severe hypertension, persistent uncontrolled diabetes, oxygen-dependent lung disease, chronic liver disease, or HIV infection.
* Patients must not have had other malignancies other than prostate cancer in the past 5 years, but cured basal cell or squamous cell skin cancers can be enrolled.
* Patients with mental illness, mental disability or inability to give informed consent are not eligible.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Time to PSA progression progression | up to 2 years
  PSA progression is defined as elevated PSA levels(≥2ng/ml) for no less than 2 measurements at least 1 week apart.
Time to Radiographic progression | up to 2 years
  Radiographic progression is defined as newly discovered soft tissue metastasis according to the RECIST 1.1 or at least 2 bone lesions.

SECONDARY OUTCOMES:
rPFS (radiographic progression free survival) | up to 2 years
  The time of radiographic progression free survival
Time to castration resistance | up to 2 years
  The time to castration resistance
Time to PSA remission (≥50%) and time to PSA remission (≥90%) | up to 2 years
  Time to the point when PSA drop to below 50% initial PSA level. Time to the point when PSA drop to below 10% initial PSA level.
Time to new anti-cancer treatment | up to 2 years
  Time to the point when onther anti-cancer treatment is necessary

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, MD, Principal Investigator — Nanjing Drum Tower Hospital, affiliated to medical school of Nanjing University
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No